CLINICAL TRIAL: NCT06027528
Title: Evaluation of Socket Preservation Using Autogenous Dentine Graft With Or Without Autologous Fibrin Glue: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Socket Preservation Using Autogenous Dentine Graft With Or Without Autologous Fibrin Glue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Islam Mohamed Sherif, Teaching assistant in periodontology department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22623
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Unrestorable Dentition
Keywords: socket preservation; alveolar ridge preservation; dentin graft; autologous fibrin glue; sticky dentin; sticky graft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dentin graft mixed with autologous fibrin glue (Experimental): extracted tooth will be grinded into small particles to form dentin graft that will be mixed with autologous fibrin glue to be grafted in the extracted socket
  Interventions: Procedure: dentin graft mixed with autologous fibrin glue
- dentin graft (Active Comparator): extracted tooth will be grafted in the extracted socket
  Interventions: Procedure: dentin graft

INTERVENTIONS:
Procedure: dentin graft mixed with autologous fibrin glue — extracted tooth will be grinded into small particles to form dentin graft that will be mixed with autologous fibrin glue to be grafted in the extracted socket using centrifuge
  Arms: dentin graft mixed with autologous fibrin glue
Procedure: dentin graft — extracted tooth will be grafted in the socket
  Arms: dentin graft

SUMMARY:
* The aim of this interventional study is to investigate the dimensional changes in buccolingual alveolar ridge width in socket preservation using sticky dentin vs dentin graft alone
* The main question: is dentin graft mixed with autologous fibrin glue has better dimensional changes than using dentin graft alone ?
* outcomes: Change in buccolingual alveolar ridge width as well as apico-coronal alveolar ridge height

DETAILED DESCRIPTION:
* Aim of the study: The aim of this study is to investigate the dimensional changes in buccolingual alveolar ridge width. As well as the apico-coronal alveolar ridge height following tooth extraction when using sticky grafts combined with demineralized dentin grafts for socket preservation.
* Research Procedure in brief:

This study will be carried out on patients enrolled from the Outpatient Clinic of Oral Medicine and Periodontology department, Faculty of Dentistry, Cairo University. *operative procedure: Before tooth extraction, probing depths (PD), gingival recession (GR), and bleeding on probing (BOP) will be assessed at six sites (mid-facial, mesio-facial, disto-facial, mid-palatal, mesio-palatal, and disto-palatal) around the tooth to be extracted and on the adjacent teeth to verify their periodontal status. Local anesthesia will be administered by infiltration to achieve the necessary anesthesia to allow extraction of the indicated tooth. Flapless atraumatic extraction will be done. Extracted teeth will be cleaned from periodontal ligaments, cementum, soft tissue attachment, caries or restorations (if present), using a high-speed stone. The pulp chamber will be cleaned with sterile endodontic files. Then, teeth will be grinded to fine particles.

The particles prepared will be immersed tooth in alcohol for 10 min for disinfection, then washed twice in saline and dried using sterile gauze.

Then the dentine graft particles will be prepared by demineralization of tooth particles in 0.6N hydrochloric acid for 30 min to achieve demineralization then washed twice in saline and dried with sterile gauze

Then the patient will be randomly assigned to one of the treatment groups:

In group 1 (control group) Demineralized dentine graft will be placed in the socket.

In group 2 (test group):

Sticky graft preparation will be done as follows:

1. Small amount of patient's venous blood (8-10cc) is drawn via venipuncture, and the blood is placed into non-coated vacutainers to obtain autologous fibrin glue (AFG), which will make sticky graft.
2. The blood in the test tubes is centrifuged at 2700-3000 rpm for 2-3 mins.
3. The upper autologous fibrin glue is obtained with syringe and mixed with particulate of dentine graft and allows for 5-10 minutes for polymerization in order to produce sticky graft.
4. The prepared sticky dentin graft will then be inserted in the socket.

   * Post operative radiograph:

Cone beam CT will be taken post surgically to measure the buccolingual dimension in the same day of the surgery.

*Post-surgical procedure: (six months after socket preservation) Another Cone beam CT will be taken to measure the outcomes by superimposition of the 2 CBCT

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients ≥18 years old
* Nonsmoker
* Teeth with root fracture, teeth with failed endodontic therapy or advanced caries
* Intact extraction socket with no dehiscence or fenestration.

Exclusion Criteria:

* Patients with systemic diseases.
* Patients with dehiscence or fenestrations
* Patients with presence or history of osteonecrosis of the jaws, with use of bisphosphonates, exposure to head and neck radiation, chemotherapy.
* Patients with large distinct pre-apical pathology
* Smokers of more than 10 cigarettes a day or equivalent to cigarettes
* Breastfeeding or pregnant women
* Patients without availability to attend follow-up visits or patients rejecting to sign the informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in buccolingual alveolar ridge width dimensions immediately after tooth extraction (baseline) and ≥ 6 months after (follow-up). | 6 month
  superimposition of the 2 CBCT and using Scans which will be exported as DICOM format to 3D viewer software

SECONDARY OUTCOMES:
changes in apico-coronal alveolar ridge height immediately after tooth extraction and 6 months after | 6 months
  superimposition of the 2 CBCT and using Scans which will be exported as DICOM format to 3D viewer software

CONTACTS AND LOCATIONS:
Overall Officials: Amr Zahran, Professor, Study Director — Cairo University